CLINICAL TRIAL: NCT03325192
Title: A Randomized, Double Blinded, Controlled Trial of a Rapid Pleurodesis Protocol After Indwelling Pleural Catheter Placement for Malignant Pleural Effusions
Brief Title: Rapid Pleurodesis Through an Indwelling Pleural Catheter
Acronym: RAPID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kevin Ma, MD, Assistant Professor of Clinical Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 827688
Record Dates: First submitted 2017-10-24; First posted 2017-10-30 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Pleural Effusion, Malignant; Pleurodesis; Pleural Diseases
Keywords: Indwelling Pleural Catheter; Pleurodesis; Iodopovidone; Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant; Pleural Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled, Double Blinded, Parallel Design, Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subject assignment will be done using randomly generated assignment tables based on stratification by tumor type (Lung, Breast, Other) and assigned 1:1 using random permuted blocks of 4.
  Subjects will be blinded to their group assignment to minimize bias on follow up surveys.
  Physicians evaluating the patient during the initial visit and on subsequent postprocedure followup will be blinded to subject assignment. The provider responsible for placement of the catheter and delivery of the pleurodesis agent or placebo will not be involved in post procedure followup care
  All treatment physicians will follow prespecified protocols in deciding on adequate pleurodesis and timing of IPC removal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Placebo Comparator): Subjects in this arm will receive placebo only (100mL of normal saline) into the pleural space delivered via the newly placed tunneled intrapleural catheter
  Interventions: Other: Placebo
- Rapid pleurodesis protocol (Experimental): Subjects in this arm will receive the chemical pleurodesing agent of 10% iodopovidone solution delivered to the pleural space via the newly placed tunneled intrapleural catheter
  Interventions: Drug: Rapid pleurodesis protocol

INTERVENTIONS:
Drug: Rapid pleurodesis protocol — * The pleural space will be evacuated completely through the newly placed IPC
  * 20mL of 10% iodopovidone and 80mL of normal saline will be instilled into the pleural space
  * The patient will be transferred to the recovery unit
  * Two hours after instillation the pleural space will be drained
  * After recovery from anesthesia and complete drainage of the pleurodesis mix, the subject will be discharged
  * Subjects will be asked to drain their effusion on a daily basis for the next 7 days and then on an every other day basis.
  Other Names: iodine pleurodesis
  Arms: Rapid pleurodesis protocol
Other: Placebo — * The pleural space will be evacuated completely through the newly placed IPC
  * Only placebo (normal saline) will be instilled into the pleural space
  * The patient will be transferred to the recovery unit
  * Two hours after instillation the pleural space will be drained
  * After recovery from anesthesia and complete drainage of the pleurodesis mix, the subject will be discharged
  * Subjects will be asked to drain their effusion on a daily basis for the next 7 days and then on an every other day basis.
  Arms: Standard of care

SUMMARY:
The primary objective of the study is to evaluate whether the use of a rapid pleurodesis protocol using 10% iodopovidone immediately after tunneled pleural catheter placement improves time to IPC removal compared to patients who receive an IPC alone.

DETAILED DESCRIPTION:
Patients will be screened throughout the year as part of the clinical referral process to the Interventional Pulmonology service at the Hospital of the University of Pennsylvania for the management of a malignant pleural effusion. Patients eligible for inclusion based on the clinical evaluation will be approached for enrollment. Written consent will be obtained. Patients will subsequently undergo placement of a IPC under MAC as per standard clinical practice followed by complete drainage of the pleural space. Patients randomized to the rapid pleurodesis protocol arm will received 20mL of 10% iodopovidone mixed with 80mL of normal saline instilled intrapleurally through the IPC. Patients randomized to the standard of care arm will have 100mL of normal saline (placebo) instilled intrapleurally through the IPC. The mixture will be allowed to dwell for 2 hours and then completely evacuated through the IPC and the patient will be discharged home.

After discharge, all patients will continue to drain their IPC on a daily basis for 7 days. Following this, all patients will continue to drain their IPC on an every-other-day basis until total IPC output is less than 50ml per session over 3 consecutive sessions. At which point they will be asked to undergo a clamp trial of no drainage for 7 days followed by a reattempt at drainage. Patients without return of symptoms over those 7 days and minimal drainage afterwards (<50ml) will be seen in the office for possible IPC removal. Patients with return of symptoms during those 7 days or more than minimal drainage afterwards (>50mL) will be asked to continue drainage until total IPC output is again less than 50mL per session over 3 sessions.

After a passed clamp trial, patients will be evaluated in the office with a bedside ultrasound to assess for pleural apposition in 5 of 6 designated points and the absence of pleural effusions. If all criteria are met, the IPC is removed. If there is evidence of residual effusion, continued drainage will be advised.

All patients will be evaluated in the office on day 7, day 14, day 30, day 60 and day 90 after IPC placement. On each visit they will be assessed for pleural apposition with ultrasound. At day 30, 60, and 90 all patients will receive a global health related questionnaire (EORTC QLQ30) and a symptom questionnaire. At 90 days, complications rate will be assessed for the entire study period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MPE as defined by

   1. A diagnosis a pleural effusion in the setting of known malignancy. AND
   2. Confirmed malignant involvement of the pleural space by fluid cytology or pleural biopsy. OR
   3. Evidence of pleural disease on radiographic imaging. OR
   4. A recurrent effusion with no other identifiable cause after thorough workup.
2. Symptomatic from the pleural effusions (shortness of breath, cough, or chest pain)
3. Prior thoracentesis with post procedure symptomatic relief
4. Recurrence of symptoms with re-accumulation of pleural effusion
5. Lung re-expansion after thoracentesis on chest imaging within last 30 days

Exclusion Criteria:

1. Malignant pleural effusion due to a hematologic malignancy
2. ECOG >4
3. Any history of trapped lung
4. Prior attempted pleurodesis on the affected site
5. Age <18
6. Pregnant or lactating
7. Known allergy to iodopovidone (Betadine)
8. Unable or unwilling to provide consent
9. Uncorrectable coagulopathy (INR > 1.5, aPTT > 1.5 x the upper limit of normal) or thrombocytopenia (< 50,000)
10. Anatomic contraindication to IPC (overlying skin abnormalities)
11. Unable or unwilling to care for IPC and adhere to drainage protocol
12. Need for bilateral IPC placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Time to catheter removal | 90 days
  Time to IPC removal will be measured in days from the day of IPC placement to the day of IPC removal after meeting removal criteria as listed above.

SECONDARY OUTCOMES:
Change in Global Health Related Quality of Life | 30 days, 60 days, and 90 days after catheter placement
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQC30) will be used to assess global health-related quality of life. This is a 30-item questionnaire validated for use in patients with cancer. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Change in symptoms of pain and breathlessness | 30 days, 60 days, and 90 days after catheter placement
  We will use a 5 point Likert scale (5PLS) that has been created for the trial. Patients will be asked to indicate their degree of shortness of breath or chest pain during sitting, walking and lying down/sleeping on that specific day. Thus, a total of 6 scales will be utilized. Point 1 will be described as "no shortness of breath" or "no chest pain." Point 2 will be described as "mild shortness of breath" or "mild chest pain." Point 3 will be described as "moderate shortness of breath" or "moderate chest pain." Point 4 will be described as "severe shortness of breath" or "severe chest pain." Point 5 will be described as "Worst shortness of breath possible" or "Worst chest pain possible."
Time to return of clinically significant pleural effusion | 90 days
  This will be measured in days from the day of IPC removal to the day of return of a clinically significant pleural effusion in the same hemithorax that originally required IPC placement. A clinically significant reaccumulation of pleural fluid will be defined as an effusion with a maximum fluid depth greater than 25% of the AP window on chest CT or 1cm thoracic ultrasound along the lateral 1/3 of the thorax that is associated with shortness of breath or chest pain
Rate of successful pleurodesis at 90 days | 90 days
  Successful pleurodesis will be defined as removal of the IPC with no clinically significant reaccumulation of pleural fluid as evaluated by chest CT or thoracic ultrasound. A clinically significant reaccumulation of pleural fluid will be defined as an effusion with a maximum fluid depth greater than 25% of the AP window on chest CT or 1cm thoracic ultrasound along the lateral 1/3 of the thorax that is associated with shortness of breath or chest pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Ma, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antunes G, Neville E, Duffy J, Ali N; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of malignant pleural effusions. Thorax. 2003 May;58 Suppl 2(Suppl 2):ii29-38. doi: 10.1136/thorax.58.suppl_2.ii29. No abstract available. PMID 12728148
- [Background] American Thoracic Society. Management of malignant pleural effusions. Am J Respir Crit Care Med. 2000 Nov;162(5):1987-2001. doi: 10.1164/ajrccm.162.5.ats8-00. No abstract available. PMID 11069845
- [Background] Davies HE, Mishra EK, Kahan BC, Wrightson JM, Stanton AE, Guhan A, Davies CW, Grayez J, Harrison R, Prasad A, Crosthwaite N, Lee YC, Davies RJ, Miller RF, Rahman NM. Effect of an indwelling pleural catheter vs chest tube and talc pleurodesis for relieving dyspnea in patients with malignant pleural effusion: the TIME2 randomized controlled trial. JAMA. 2012 Jun 13;307(22):2383-9. doi: 10.1001/jama.2012.5535. PMID 22610520
- [Background] Roberts ME, Neville E, Berrisford RG, Antunes G, Ali NJ; BTS Pleural Disease Guideline Group. Management of a malignant pleural effusion: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii32-40. doi: 10.1136/thx.2010.136994. No abstract available. PMID 20696691
- [Background] Wahidi MM, Reddy C, Yarmus L, Feller-Kopman D, Musani A, Shepherd RW, Lee H, Bechara R, Lamb C, Shofer S, Mahmood K, Michaud G, Puchalski J, Rafeq S, Cattaneo SM, Mullon J, Leh S, Mayse M, Thomas SM, Peterson B, Light RW. Randomized Trial of Pleural Fluid Drainage Frequency in Patients with Malignant Pleural Effusions. The ASAP Trial. Am J Respir Crit Care Med. 2017 Apr 15;195(8):1050-1057. doi: 10.1164/rccm.201607-1404OC. PMID 27898215
- [Background] Lui MM, Thomas R, Lee YC. Complications of indwelling pleural catheter use and their management. BMJ Open Respir Res. 2016 Feb 5;3(1):e000123. doi: 10.1136/bmjresp-2015-000123. eCollection 2016. PMID 26870384
- [Background] Reddy C, Ernst A, Lamb C, Feller-Kopman D. Rapid pleurodesis for malignant pleural effusions: a pilot study. Chest. 2011 Jun;139(6):1419-1423. doi: 10.1378/chest.10-1868. Epub 2010 Oct 7. PMID 20930006
- [Background] Krochmal R, Reddy C, Yarmus L, Desai NR, Feller-Kopman D, Lee HJ. Patient evaluation for rapid pleurodesis of malignant pleural effusions. J Thorac Dis. 2016 Sep;8(9):2538-2543. doi: 10.21037/jtd.2016.08.55. PMID 27747006
- [Background] Boujaoude Z, Bartter T, Abboud M, Pratter M, Abouzgheib W. Pleuroscopic Pleurodesis Combined With Tunneled Pleural Catheter for Management of Malignant Pleural Effusion: A Prospective Observational Study. J Bronchology Interv Pulmonol. 2015 Jul;22(3):237-43. doi: 10.1097/LBR.0000000000000186. PMID 26165894
- [Background] Ahmed L, Ip H, Rao D, Patel N, Noorzad F. Talc pleurodesis through indwelling pleural catheters for malignant pleural effusions: retrospective case series of a novel clinical pathway. Chest. 2014 Dec;146(6):e190-e194. doi: 10.1378/chest.14-0394. PMID 25451360
- [Background] King MT. The interpretation of scores from the EORTC quality of life questionnaire QLQ-C30. Qual Life Res. 1996 Dec;5(6):555-67. doi: 10.1007/BF00439229. PMID 8993101
- [Background] Sivakumar P, Douiri A, West A, Rao D, Warwick G, Chen T, Ahmed L. OPTIMUM: a protocol for a multicentre randomised controlled trial comparing Out Patient Talc slurry via Indwelling pleural catheter for Malignant pleural effusion vs Usual inpatient Management. BMJ Open. 2016 Oct 18;6(10):e012795. doi: 10.1136/bmjopen-2016-012795. PMID 27798020
- [Background] Neto JD, de Oliveira SF, Vianna SP, Terra RM. Efficacy and safety of iodopovidone pleurodesis in malignant pleural effusions. Respirology. 2010 Jan;15(1):115-8. doi: 10.1111/j.1440-1843.2009.01663.x. Epub 2009 Nov 23. PMID 19947987
- [Background] Agarwal R, Paul AS, Aggarwal AN, Gupta D, Jindal SK. A randomized controlled trial of the efficacy of cosmetic talc compared with iodopovidone for chemical pleurodesis. Respirology. 2011 Oct;16(7):1064-9. doi: 10.1111/j.1440-1843.2011.01999.x. PMID 21605278
- [Background] Olivares-Torres CA, Laniado-Laborin R, Chavez-Garcia C, Leon-Gastelum C, Reyes-Escamilla A, Light RW. Iodopovidone pleurodesis for recurrent pleural effusions. Chest. 2002 Aug;122(2):581-3. doi: 10.1378/chest.122.2.581. PMID 12171835
- [Background] Godazandeh G, Qasemi NH, Saghafi M, Mortazian M, Tayebi P. Pleurodesis with povidone-iodine, as an effective procedure in management of patients with malignant pleural effusion. J Thorac Dis. 2013 Apr;5(2):141-4. doi: 10.3978/j.issn.2072-1439.2013.02.02. PMID 23585939
- [Background] Agarwal R, Aggarwal AN, Gupta D, Jindal SK. Efficacy and safety of iodopovidone in chemical pleurodesis: a meta-analysis of observational studies. Respir Med. 2006 Nov;100(11):2043-7. doi: 10.1016/j.rmed.2006.02.009. Epub 2006 Mar 30. PMID 16574389